CLINICAL TRIAL: NCT02778022
Title: Child Adult Relationship Enhancement in Pediatric Primary Care Parenting Group to Reduce Child Behavior Problems
Acronym: PriCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Oscar G. & Elsa S. Mayer Family Foundation (Unknown); The Pew Charitable Trusts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-012604
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Child Behavior Disorders
Keywords: Child behavior disorders; Parent child relationship; Primary care
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study team member who will administer the follow-up study interviews will remain blinded to the group status throughout the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate PriCARE (Experimental): Parent-child dyads assigned to the immediate PriCARE group will receive the PriCARE intervention as soon as possible plus usual treatment. The intervention will last approximately 6-8 weeks. Each group will have approximately 4-13 participants and 2 facilitators and will meet 6 times for 1-2 hours per session. Parents are expected to practice the skills they learn with their children between sessions.
  Interventions: Behavioral: PriCARE
- Delayed PriCARE (No Intervention): The delayed PriCARE group will not receive the PriCARE intervention until after their data collection for this study is complete (in 3-6 months). In addition, they will be immediately offered usual treatment. Under usual treatment, patients will be referred to a behavioral health specialist at the discretion of their pediatrician and the office social worker for additional diagnosis and treatment and/or provided with a 1-2 page informational handout on child behavior problems from the CHOP patient care manual.

INTERVENTIONS:
Behavioral: PriCARE — PriCARE is a group parent training program designed to improve child behavior, improve parent-child relationships, and decrease stress for parents. PriCARE utilizes the 3 P skills (Praise, Paraphrase and Point-out-Behavior) and includes a trauma and stress education component. The training starts with parenting skills focused on giving attention to children's positive, pro-social behaviors, while ignoring minor misbehaviors. The second phase of the training teaches techniques for giving children effective commands in order to set age-appropriate limits. We piloted PriCARE and demonstrated promising findings. The PriCARE intervention has been slightly modified from the pilot version to increase engagement and attendance.
  Other Names: Child Adult Relationship Enhancement in Pediatric Primary Care
  Arms: Immediate PriCARE

SUMMARY:
The purpose of this study is to evaluate the effectiveness of PriCARE in decreasing child behavior problems and improving parenting capacity and skills at 4 primary care clinics in Philadelphia.

DETAILED DESCRIPTION:
Child behavioral concerns are common among families served by The Children's Hospital of Philadelphia (CHOP) urban primary care centers. To address this, we developed Child Adult Relationship Enhancement Model in Primary Care Parenting Program (PriCARE), a scaled down version of Parent Child Interaction Therapy designed for urban primary care clinics. The objectives of this study are to 1) evaluate the efficacy of the modified PriCARE to decrease child behavior problems and improve parenting capacity and skills and 2) understand parents' perceptions of the efficacy of PriCARE and strategies for improving its implementation and dissemination. We will perform a randomized controlled trial (RCT) of the effectiveness of the modified PriCARE on decreasing child behavior problems and improving positive parenting among 2- to 6-year-old children with behavior problems and their parents at CHOP's urban Primary Care Centers. We intend to randomize 120 child-parent pairs (240 subjects) to receive PriCARE immediately plus usual treatment (intervention group) and 60 child-parent pairs (120 subjects) to receive PriCARE at a later time plus usual treatment (control group) for a total of 180 child-parent pairs (360 subjects). All child-parent pairs randomized to the control group will be placed on a waitlist and offered PriCARE after completion of data collection. Child behavior and parenting style will be measured at baseline (time 1), at 6-19 weeks (time 2), and at 14-27 weeks (time 3).

ELIGIBILITY:
Inclusion Criteria:

1. Parent is 18 years or older
2. Parent is English speaking
3. Child is 2-6 years old
4. Parent reports that child has a behavior problem
5. Child attends CHOP Urban Primary Care Center 6) Parental/guardian permission is provided (informed consent)

Exclusion Criteria:

1. Child has a cognitive age less than 2 years old as determined by the referring clinician
2. Child is already receiving behavioral health therapy or medication (other than medication for ADHD)

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Change in Eyberg Child Behavior Inventory (ECBI) score between baseline and time 3. | baseline (time 1), 6-19 weeks (time 2), and 14-27 weeks (time 3)
  The primary objective of this study is to determine if the modified PriCARE program decreases the intensity and frequency of behavior problems in 2- to 6-year-old children as measured by the change in ECBI score after 3-7 months compared to usual treatment for child behavior problems at CHOP's South Philadelphia Primary Care Center or Karabots Pediatric Care Center. As sub-analyses, we will determine 1) the impact of caregiver depression (as measured by the Brief Symptom Inventory, BSI) on the efficacy of PriCARE intervention to decrease behavioral problems and 2) the impact of the number of PriCARE sessions attended on the efficacy of the PriCARE intervention to decrease behavioral problems.

SECONDARY OUTCOMES:
Change in Adult Adolescent Parenting Inventory-2 (AAPI-2) score between baseline and time 3 | baseline (time 1), 6-19 weeks (time 2), and 14-27 weeks (time 3)
  We will assess the efficacy of the modified PriCARE on decreasing harsh parenting as measured by the AAPI-2.
Change in Parenting Stress Index (PSI) score between baseline and time 3 | baseline (time 1), 6-19 weeks (time 2), and 14-27 weeks (time 3)
  We will assess the efficacy of the modified PriCARE on decreasing parenting stress as measured by the PSI.
Association between the Therapeutic Attitude Inventory (TAI) score and the change in ECBI score from baseline to time 2 and 3 in the immediate PriCARE group. | 14-27 weeks (time 3)
  We will assess parents' perceptions of the efficacy of the modified PriCARE on improving parenting skills and child behavior as measured by the TAI.
Conceptual model of facilitators and barriers to participation in behavioral interventions in primary care as well as the strengths and weaknesses of the PriCARE program | 6-27 weeks
  We will conduct a qualitative interview with up to 30 parents randomized to the immediate PriCARE group to gain an understanding of how implementation and dissemination of the modified PriCARE can be improved in order to increase attendance and maximize effectiveness.
Change in The Keys to Interactive Parenting Scale (KIPS) score between baseline and time 3 | baseline (time 1) and 14-27 weeks (time 3)
  As an exploratory aim, we will pilot the use of a video observation measure of parent-child interaction (KIPS) in assessing the impact of PriCARE on parenting behaviors with a subset of subjects.

OTHER OUTCOMES:
Description of study groups | baseline
  Demographics and baseline measures of child behavior (ECBI), parent intimate partner violence (HITS), and parent depression (BSI) for the intervention and control groups will be examined to ensure randomization resulted in comparable populations.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne N Wood, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weitzman C, Wegner L; Section on Developmental and Behavioral Pediatrics; Committee on Psychosocial Aspects of Child and Family Health; Council on Early Childhood; Society for Developmental and Behavioral Pediatrics; American Academy of Pediatrics. Promoting optimal development: screening for behavioral and emotional problems. Pediatrics. 2015 Feb;135(2):384-95. doi: 10.1542/peds.2014-3716. PMID 25624375
- [Background] Bultas MW, McMillin SE, Broom MA, Zand DH. Brief, Rapid Response, Parenting Interventions Within Primary Care Settings. J Behav Health Serv Res. 2017 Oct;44(4):695-699. doi: 10.1007/s11414-015-9479-2. PMID 26289564
- [Background] Querido JG, Warner TD, Eyberg SM. Parenting styles and child behavior in African American families of preschool children. J Clin Child Adolesc Psychol. 2002 Jun;31(2):272-7. doi: 10.1207/S15374424JCCP3102_12. PMID 12056110
- [Background] Asarnow JR, Rozenman M, Wiblin J, Zeltzer L. Integrated Medical-Behavioral Care Compared With Usual Primary Care for Child and Adolescent Behavioral Health: A Meta-analysis. JAMA Pediatr. 2015 Oct;169(10):929-37. doi: 10.1001/jamapediatrics.2015.1141. PMID 26259143
- [Background] Meadows T, Valleley R, Haack MK, Thorson R, Evans J. Physician "costs" in providing behavioral health in primary care. Clin Pediatr (Phila). 2011 May;50(5):447-55. doi: 10.1177/0009922810390676. Epub 2010 Dec 30. PMID 21196418
- [Background] Ward-Zimmerman B, Cannata E. Partnering with pediatric primary care: Lessons learned through collaborative colocation. Professional Psychology: Research and Practice. 2012;43(6):596-605.
- [Background] Schuhmann EM, Foote RC, Eyberg SM, Boggs SR, Algina J. Efficacy of parent-child interaction therapy: interim report of a randomized trial with short-term maintenance. J Clin Child Psychol. 1998 Mar;27(1):34-45. doi: 10.1207/s15374424jccp2701_4. PMID 9561935
- [Background] Sherin KM, Sinacore JM, Li XQ, Zitter RE, Shakil A. HITS: a short domestic violence screening tool for use in a family practice setting. Fam Med. 1998 Jul-Aug;30(7):508-12. PMID 9669164
- [Background] Morlan KK, Tan SY. Comparison of the Brief Psychiatric Rating Scale and the Brief Symptom Inventory. J Clin Psychol. 1998 Nov;54(7):885-94. doi: 10.1002/(sici)1097-4679(199811)54:73.0.co;2-e. PMID 9811126
- [Background] Conners NA, Whiteside-Mansell L, Deere D, Ledet T, Edwards MC. Measuring the potential for child maltreatment: the reliability and validity of the Adult Adolescent Parenting Inventory--2. Child Abuse Negl. 2006 Jan;30(1):39-53. doi: 10.1016/j.chiabu.2005.08.011. Epub 2006 Jan 6. PMID 16406026
- [Background] Eyberg SM, Ross AW. Assessment of Child Behavior Problems: The Validation of a New Inventory. J Clin Child Psycho. 1978.
- [Background] Abidin RR. Parenting Stress Index. 4th ed. Lutz, FL: PAR; 2012.
- [Background] Brestan EV JJ, Rayfield AD, Eybert SM. A consumer satisfaction measure for parent-child treatments and its relation to measures of child behavior change. Behavior Therapy. 1999;30:17-30.
- [Background] Comfort M, Gordon PR. The Keys to Interactive Parenting Scale (KIPS): A practical observational assessment of parenting behavior. NHSA Dialog: A Research-To-Practice Journal for the Early Intervention Field. Vol 9(1). Alexandria, VA: National Head Start Association Research and Evaluation Department; 2006:22-48.